CLINICAL TRIAL: NCT00646256
Title: Psychoeducation in Patients With Schizophrenia: Neuropsychological Performance and Cognitive Training as Determinants of Outcome
Brief Title: Cognitive Determinants of Psychoeducation and Information in Psychoses
Acronym: COGPIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Research Foundation (Other)
Responsible Party: Prof. Dr. phil. Dipl.-Psych. Thomas Jahn, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFG Ja 680 / 4-2, 4-3
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Schizophrenia; Delusional Disorders (ICD-10)
Keywords: schizoaffective; schizotypal
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Paranoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no training (No Intervention)
- COGPACK training (Experimental)
  Interventions: Behavioral: COGPACK training, psychoeducation

INTERVENTIONS:
Behavioral: COGPACK training, psychoeducation — Bifocal psychoeducation group program (Munich Psychoses Information Program - PIP) with preceding computerbased cognitive training program (COGPACK)
  Arms: COGPACK training

SUMMARY:
The aim of the study is to examine whether the efficacy of psychoeducation in patients with schizophrenia or schizoaffective disorders is dependent on their cognitive performance level and if a preceding cognitive training can enhance the therapeutic effects of psychoeducation

DETAILED DESCRIPTION:
Schizophrenic inpatients are examined shortly after admission with a broad battery of clinical and neurological rating scales and neuropsychological tests. They are then randomized to either standard treatment (including antipsychotic medications, art and occupational therapy, psychotherapy) or to standard treatment plus daily computerbased cognitive training (COGPACK; ten 1-hour sessions over two weeks). After repetition of the broad assessment battery all patients (and some of their family members) take part in a bifocal psychoeducation group program (eight 1-hour sessions over four weeks). Specific pre-post measures are illness knowledge, self and expert ratings of adherence to treatment, insight to the illness, treatment satisfaction. The study also includes a 9-month follow-up, with number of rehospitalizations, days in hospital and psychopathology as the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* Informed consent
* German as first language or very good knowledge of German

Exclusion Criteria:

* Mental retardation
* Any serious somatic illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
illness knowledge, adherence to treatment, insight to the illness, satisfaction with treatment. 9-month follow-up: number of rehospitalizations, days in hospital | Baseline, after cognitive training, after psychoeducation, 9-month after end of psychoeducation

SECONDARY OUTCOMES:
Psychopathological status
Psychosocial rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jahn, Prof. Dr. phil. Dipl.-Psych., Principal Investigator — Klinik und Poliklinik für Psychiatrie und Psychotherapie, Klnikum rechts der Isar, Technbical Univesity Munich
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Klinikum rechts der Isar, Technical University of Munich, Munich, Germany

REFERENCES:
- [Derived] Pitschel-Walz G, Bauml J, Frobose T, Gsottschneider A, Jahn T. Do individuals with schizophrenia and a borderline intellectual disability benefit from psychoeducational groups? J Intellect Disabil. 2009 Dec;13(4):305-20. doi: 10.1177/1744629509353237. PMID 20048350